CLINICAL TRIAL: NCT06549426
Title: Treatment of ELectrographic STatus Epilepticus After Cardiopulmonary Resuscitation-2: Multicenter Randomised Clinical Trial and Health Economic Evaluation of Anti-seizure Treatment in Comatose Cardiac Arrest Patients With SE on Continuous EEG
Brief Title: Treatment of ELectroencephalographic STatus Epilepticus After Cardiopulmonary Resuscitation-2 (TELSTAR-2)
Acronym: TELSTAR-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Collaborators: Erasme University Hospital (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Principal Investigator, Jeannette Hofmeijer, prof. dr., University of Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-516068-27-01
Record Dates: First submitted 2024-08-02; First posted 2024-08-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Coma; Electrographic Status Epilepticus
MeSH Terms: conditions — Coma; Status Epilepticus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Standard care completed with stepwise anti-seizure treatment according to protocols for clinically overt status epilepticus. This consists of a stepwise approach consisting of 3 potential steps. Each next step will be taken as soon as possible (within 30 minutes of ESE first diagnosis or recurrence) if the previous step was insufficiently effective to sustainably suppress ESE.
  Interventions: Drug: anti-seizure medication + sedative agent(s)
- Control group (No Intervention): Standard care without anti-seizure treatment.

INTERVENTIONS:
Drug: anti-seizure medication + sedative agent(s) — Stepwise approach:
  1. a single dose of a parenteral benzodiazepine (lorazepam, midazolam, or diazepam) and a first parenteral anti-seizure medication (levetiracetam, valproate, or lacosamide)
  2. a second parenteral anti-seizure medication plus a first continuous parenteral sedative agent (midazolam or propofol)
  3. a second continuous parenteral sedative agent (midazolam, propofol, or ketamine)
  Arms: Intervention group

SUMMARY:
The goal of this comparative effectiveness trial is to study electrographic status epilepticus (ESE) treatment in comatose patients after cardiac arrest. The main questions the trial aims to answer are:

* Does ESE treatment improve outcome?
* What is the impact of ESE treatment on healthcare costs?

Participants in the the intervention group will receive standard care completed with anti-seizure treatment. The control group will receive standard care without anti-seizure treatment.

DETAILED DESCRIPTION:
Rationale: Around 7500 comatose patients after cardiac arrest and resuscitation are admitted to intensive care units (ICUs) in the Netherlands and Belgium, yearly. Approximately half eventually dies from severe brain injury. EEG is used as a predictor of outcome, helping decide whether life sustaining therapies should be pursued or withdrawn. EEG shows epileptiform patterns meeting criteria for electrographic status epilepticus (ESE) in up to 10% of patients, with 80-100% case fatality. With the TELSTAR-1 trial, we showed that anti-seizure treatment of unselected patients with epileptiform patterns is not associated with a better outcome. However, it remains unclear whether treatment of (possible) ESE will improve outcome, or if ESE simply represents irreversible severe brain damage, in which case such treatment will be futile. This translates into ongoing practice variation. To provide comatose cardiac arrest survivors with the best medical treatment options, while at the same time preventing unnecessary costly ICU treatment, unequivocal evidence of efficacy or futility of ESE treatment is needed.

Objectives: It is the primary objective to study whether ESE treatment improves outcome of comatose patients after cardiac arrest. It is the secondary objective to study the impact on healthcare costs of ESE treatment.

Main trial endpoints: The primary outcome measure will be functional recovery expressed as the score on the extended Glasgow Outcome Scale (eGOS) at six months after cardiac arrest. The primary effect parameter will be the common odds ratio for any shift towards a better outcome in the intervention group, analyzed by multivariable ordinal logistic regression.

Secondary trial endpoints: Secondary outcome measures include data on quality of life, cognitive functioning, and the use of resources. Cost-effectiveness will be assessed, separately for Belgium and for the Netherlands, adhering to 'KCE' and 'Zorginstituut' guidelines for pharmaco-economic evaluations, respectively.

Trial design: This will be a comparative effectiveness study, comparing two standard treatment regimens. We will conduct a prospective multicentre trial with randomized treatment allocation, open label treatment, and blinded endpoint assessment on twenty intensive care units in the Netherlands and Belgium.

Trial population: The study population consists of adult comatose patients after out of hospital cardiac arrest and successful cardiopulmonary resuscitation, admitted on the intensive care unit of any of the participating centres, with ESE on continuous EEG. Continuous EEG is part of standard care in all participating hospitals. For the definition of ESE, we adhere to international consensus criteria.

Interventions: Treatment in the intervention group will consist of standard care completed with anti-seizure treatment according to protocols for clinically overt status epilepticus with the goal of definitive seizure suppression. This consists of a stepwise approach, step 1 being a single dose of a parenteral benzodiazepine (lorazepam, midazolam, or diazepam) and a first parenteral anti-seizure medication (levetiracetam, valproate, or lacosamide), step 2, a second parenteral anti-seizure medication plus a first continuous parenteral sedative agent (midazolam or propofol), and step 3, a second continuous parenteral sedative agent (midazolam, propofol, or ketamine). Each next step will be taken as soon as possible (within 30 minutes) if the previous step was insufficiently effective to suppress ESE. The control group will receive standard care without anti-seizure treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Coma (Glasgow Coma Scale score ≤ 8) after out of hospital cardiac arrest and resuscitation
2. Age ≥ 18 years
3. Continuous EEG with at least eight electrodes started < 24h after return of spontaneous circulation (ROSC)
4. ESE or possible ESE according to the Salzburg and ACNS criteria
5. Possibility to start treatment within three hours after detection of ESE

Exclusion Criteria:

1. Known history of another medical condition with limited life expectancy (< six months)
2. Any progressive brain illness, such as a brain tumor or neurodegenerative disease
3. Pre-admission Glasgow Outcome Scale score of 3 or lower
4. Reason other than the neurological condition to withdraw treatment
5. EEG background activity prior to the emergence of ESE indicative of extensive irreversible anoxic brain injury
6. Follow-up impossible due to logistic reasons, for example not living in the Netherlands or Belgium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
score on the extended Glasgow Outcome Scale (eGOS) | 6 months after cardiac arrest
  eGOS is an 8-points ordinal scale of functional recovery with possible scores ranging from 0 to 6. A higher score indicates better functional recovery

SECONDARY OUTCOMES:
quality adjusted life years (QALYs) | 12 months after cardiac arrest
  this is a measure of cost-effectiveness

OTHER OUTCOMES:
survival in months | 12 months after cardiac arrest
  this is a measure of survival
death (any cause), pneumonia, sepsis (according to sepsis 3 criteria), bleeding (any cause), cardiac arrhythmia (any associated with hemodynamic compromise), new cardiac arrest, or thrombopenia | 12 months after cardiac arrest
  these are safety outcomes
score on the Rankin Scale (mRS) | 6 and 12 months after cardiac arrest
  mRS is a 6-point ordinal functional recovery scale with possible scores ranging from 1 to 6. A lower score indicates better functional recovery.
score on the cerebral performance categories (CPC) | 6 and 12 months after cardiac arrest
  COC is a 5-point ordinal functional recovery scale with possible scores ranging from 1 to 5. A lower score indicates better functional recovery.
score on Montreal Cognitive Assessment telephone version | 6 months after cardiac arrest
  MoCA is a screening instrument to quantify overall cognitive functioning. Scores range from 0 to 30 with higher scores indicating better cognitive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Hofmeijer, MD, Principal Investigator — University of Twente
Locations (20):
- Belgium (8):
  - Centre Hospitalier Universitaire Saint-Pierre, Brussels
  - Hôpital Universitaire de Bruxelles, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Centre Hospitalier Universitaire Marie Curie, Charleroi
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Chrétien - MontLégia, Liège
  - Centre Hospitalier Universitaire Sart-Tilmant, Liège
- Netherlands (12):
  - Amsterdam University Medical Center, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Catharina Hospital, Eindhoven
  - Medical Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - St. Antonius Hospital, Nieuwegein
  - Canisius Wilhelmina Hospital, Nijmegen
  - Radboud University Medical Center, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - Maasstad Hospital, Rotterdam
  - VieCuri Medical Center, Venlo

IPD SHARING:
Plan to Share IPD: No